CLINICAL TRIAL: NCT04462575
Title: Reconstruction of Horizontally Deficient Atrophic Maxillary Ridges Using Mandibular Blocks With and Without Coverage Using Collagen Membrane
Brief Title: Reconstruction of Atrophic Maxillary Ridges Using Mandibular Blocks With and Without Coverage Using Collagen Membrane
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohannad Ahmed Ismail, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OMFS - (3-3-14)
Record Dates: First submitted 2020-06-28; First posted 2020-07-08 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Bone Augmentation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Onlay bone block covered using collagen membrane (Experimental): The onlay bone block (harvested from mandibular intra oral sites) on top of a mixture of particulate autogenous bone and particulate xenogenic bone (assembly going to be fixed by at least 2 micro screws of diameter 1.5 mms and length 13 mms, to avoid micro movements of onlay bone block) covered by collagen membrane, stabilized by resorbable suture and fixed by tacs.
  Interventions: Procedure: Onlay bone block covered using collagen membrane
- Onlay bone block without collagen membrane (Active Comparator): The onlay bone block (harvested from mandibular intra oral sites) on top of a mixture of particulate autogenous bone and particulate xenogenic bone (assembly going to be fixed by at least 2 micro screws of diameter 1.5 mms and length 13 mms, to avoid micro movements of onlay bone block).
  Interventions: Procedure: Onlay bone block without collagen membrane

INTERVENTIONS:
Procedure: Onlay bone block covered using collagen membrane — The ratio is 40% of xenogenic bone particles (low resorption rate) to 60% of autogenous bone particles (contains viable cells) to be placed in recipient decorticated site and covered by onlay bone block..
  Arms: Onlay bone block covered using collagen membrane
Procedure: Onlay bone block without collagen membrane — Onlay bone block without collagen membrane
  Arms: Onlay bone block without collagen membrane

SUMMARY:
Is the use of collagen membrane on top of particulate bone mixture covered by onlay bone block in Maxilla better than the use of mixture of particulate bone covered by onlay bone block without the use of collagen membrane, in terms of bone quality and bone quantity?

DETAILED DESCRIPTION:
Soft tissue dehiscence could result due to flap irritation as a result of, closure under tension, intraoperative or postoperative recipient site infection, postoperative edema, which in turns compromises stability of onlay bone blocks thus osseintegration of bone block. Any attempt of bone recontouring and resuturing fails since there is no vascular bed. Ideal requirements of barrier membranes are, they should be biological compatible, they must act as a barrier membrane, unwanted fibroblasts should be hindered from entrance while allowing diffusion of nutrients, tissue integration (biological adhesion), tissues should be able to grow into the membrane but not through it. Space maintainer, it should be sufficiently stiff, so as not to collapse into the underlying particulate bone under the pressure of soft tissue and it should be ease in its manipulation, adaptation and handling, as for example, collagen membrane. Some types of collagen membrane, contain some degrees of stretchability.

ELIGIBILITY:
Inclusion Criteria:

* Patients with maxillary residual alveolar bone height not less than 8 mm.
* Alveolar bone width from less than or equal 5 mm.
* Both sexes.
* At least missing single tooth.
* Previous Failed Implants.
* Previous Failed Grafting.

Exclusion Criteria:

* Heavy smokers more than 10 cigarettes per day.
* Patients with alcohol abuse
* Patients with narcotic abuse.
* Patients with bone disease that may affect normal healing, example; hyperparathyroidism.
* Patients had radiotherapy and chemotherapy in head and neck.
* Patients had neoplasms in sites to be grafted. 18
* Patients with Metabolic diseases uncontrolled diabetic patients, Glycated hemoglobin (Hb A1c) more than 7 mg\dl.
* Pregnant females.
* Patients with Para functional habits, apprehensive and non-cooperative.
* Bone pathology related to the site to be grafted.
* Psychological problems, stress situation (socially or professionally), emotional instability, and unrealistic patients' expectations.
* Intraoral soft and hard tissue pathology.
* Systemic condition that contraindicate implant placement.
* Under the age of 18 years.

Ages: 18 Years to 46 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Quantity of bone gain. | after 4 months from ridge augmentation.
  Measured using linear measurements from Cone Beam Computed Tomography (CBCT) in millimeters (mm).

SECONDARY OUTCOMES:
Bone Quality. | after 4 months from ridge augmentation.
  Measured using Image Analyser Computer System using Histomorphometric method (area percent micrometer square) and optical density

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hammerle CH, Jung RE. Bone augmentation by means of barrier membranes. Periodontol 2000. 2003;33:36-53. doi: 10.1046/j.0906-6713.2003.03304.x. No abstract available. PMID 12950840
- [Background] Cash and Alex: 20 years of guided bone regeneration in implant dentistry, 2nd ed. (2009).
- [Background] Urban IA, Nagursky H, Lozada JL. Horizontal ridge augmentation with a resorbable membrane and particulated autogenous bone with or without anorganic bovine bone-derived mineral: a prospective case series in 22 patients. Int J Oral Maxillofac Implants. 2011 Mar-Apr;26(2):404-14. PMID 21483894
- [Background] Urban IA, Nagursky H, Lozada JL, Nagy K. Horizontal ridge augmentation with a collagen membrane and a combination of particulated autogenous bone and anorganic bovine bone-derived mineral: a prospective case series in 25 patients. Int J Periodontics Restorative Dent. 2013 May-Jun;33(3):299-307. doi: 10.11607/prd.1407. PMID 23593623
- [Background] Pellegrino G, Lizio G, Corinaldesi G, Marchetti C. Titanium Mesh Technique in Rehabilitation of Totally Edentulous Atrophic Maxillae: A Retrospective Case Series. J Periodontol. 2016 May;87(5):519-28. doi: 10.1902/jop.2016.150432. Epub 2016 Jan 12. PMID 26759078
- [Background] Polis-Yanes C, Cadenas-Sebastian C, Gual-Vaques P, Ayuso-Montero R, Mari-Roig A, Lopez-Lopez J. Guided Bone Regeneration of an Atrophic Maxilla Using Heterologous Cortical Lamina. Case Rep Dent. 2019 Jun 11;2019:5216362. doi: 10.1155/2019/5216362. eCollection 2019. PMID 31308978
- [Background] Jensen J, Sindet-Pedersen S. Autogenous mandibular bone grafts and osseointegrated implants for reconstruction of the severely atrophied maxilla: a preliminary report. J Oral Maxillofac Surg. 1991 Dec;49(12):1277-87. doi: 10.1016/0278-2391(91)90303-4. PMID 1955919
- [Background] Misch CM. Comparison of intraoral donor sites for onlay grafting prior to implant placement. Int J Oral Maxillofac Implants. 1997 Nov-Dec;12(6):767-76. PMID 9425757
- [Background] Montazem A, Valauri DV, St-Hilaire H, Buchbinder D. The mandibular symphysis as a donor site in maxillofacial bone grafting: a quantitative anatomic study. J Oral Maxillofac Surg. 2000 Dec;58(12):1368-71. doi: 10.1053/joms.2000.18268. PMID 11117684
- [Background] Gungormus M, Yavuz MS. The ascending ramus of the mandible as a donor site in maxillofacial bone grafting. J Oral Maxillofac Surg. 2002 Nov;60(11):1316-8. doi: 10.1053/joms.2002.35731. PMID 12420267
- [Background] Clavero J, Lundgren S. Ramus or chin grafts for maxillary sinus inlay and local onlay augmentation: comparison of donor site morbidity and complications. Clin Implant Dent Relat Res. 2003;5(3):154-60. doi: 10.1111/j.1708-8208.2003.tb00197.x. PMID 14575631
- [Background] Pourabbas R, Nezafati S. Clinical results of localized alveolar ridge augmentation with bone grafts harvested from symphysis in comparison with ramus. J Dent Res Dent Clin Dent Prospects. 2007 Spring;1(1):7-12. doi: 10.5681/joddd.2007.002. Epub 2007 Jun 10. PMID 23277827
- [Background] Acocella A, Bertolai R, Colafranceschi M, Sacco R. Clinical, histological and histomorphometric evaluation of the healing of mandibular ramus bone block grafts for alveolar ridge augmentation before implant placement. J Craniomaxillofac Surg. 2010 Apr;38(3):222-30. doi: 10.1016/j.jcms.2009.07.004. Epub 2009 Aug 3. PMID 19648020
- [Background] Spin-Neto R, Landazuri Del Barrio RA, Pereira LA, Marcantonio RA, Marcantonio E, Marcantonio E Jr. Clinical similarities and histological diversity comparing fresh frozen onlay bone blocks allografts and autografts in human maxillary reconstruction. Clin Implant Dent Relat Res. 2013 Aug;15(4):490-7. doi: 10.1111/j.1708-8208.2011.00382.x. Epub 2011 Aug 11. PMID 21834864
- [Background] Acocella A, Bertolai R, Ellis E 3rd, Nissan J, Sacco R. Maxillary alveolar ridge reconstruction with monocortical fresh-frozen bone blocks: a clinical, histological and histomorphometric study. J Craniomaxillofac Surg. 2012 Sep;40(6):525-33. doi: 10.1016/j.jcms.2011.09.004. Epub 2011 Nov 9. PMID 22075326
- [Background] Dasmah A, Thor A, Ekestubbe A, Sennerby L, Rasmusson L. Particulate vs. block bone grafts: three-dimensional changes in graft volume after reconstruction of the atrophic maxilla, a 2-year radiographic follow-up. J Craniomaxillofac Surg. 2012 Dec;40(8):654-9. doi: 10.1016/j.jcms.2011.10.032. Epub 2011 Dec 3. PMID 22137760
- [Background] AlGhamdi AS. Post-surgical complications of symphyseal block graft with and without soft tissue grafting. Saudi Med J. 2013 Jun;34(6):609-15. PMID 23756926
- [Background] Hernandez-Alfaro F, Sancho-Puchades M, Guijarro-Martinez R. Total reconstruction of the atrophic maxilla with intraoral bone grafts and biomaterials: a prospective clinical study with cone beam computed tomography validation. Int J Oral Maxillofac Implants. 2013 Jan-Feb;28(1):241-51. doi: 10.11607/jomi.2405. PMID 23377071
- [Background] Monje A, Monje F, Chan HL, Suarez F, Villanueva-Alcojol L, Garcia-Nogales A, Wang HL. Comparison of microstructures between block grafts from the mandibular ramus and calvarium for horizontal bone augmentation of the maxilla: a case series study. Int J Periodontics Restorative Dent. 2013 Nov-Dec;33(6):e153-61. doi: 10.11607/prd.1664. PMID 24116370
- [Background] Aloy-Prosper A, Penarrocha-Oltra D, Penarrocha-Diago M, Penarrocha-Diago M. The outcome of intraoral onlay block bone grafts on alveolar ridge augmentations: a systematic review. Med Oral Patol Oral Cir Bucal. 2015 Mar 1;20(2):e251-8. doi: 10.4317/medoral.20194. PMID 25662543
- [Background] Reininger D, Cobo-Vazquez C, Monteserin-Matesanz M, Lopez-Quiles J. Complications in the use of the mandibular body, ramus and symphysis as donor sites in bone graft surgery. A systematic review. Med Oral Patol Oral Cir Bucal. 2016 Mar 1;21(2):e241-9. doi: 10.4317/medoral.20938. PMID 26827063
- [Background] Khoury F: Augmentation of severe bony defects with intraoral bone grafts: biological approach and long-term results J Oral Maxillo Fac Surg 2017Volume 46, Supplement 1, Pages 26-27.
- [Background] Claudino M, Julio C L, Luis E M, Bernardo M, Fernando G, tomographic evaluation of atrophic maxilla rehabilitated with autogenous and xenogeneic block grafts. Journal of Research in Dentistry 2017, 4(4):112-117.
- [Derived] Ismail M, Shawky M, Fattouh H, Mounir M, El Moshy S, Askar N, Atef M. Horizontal Maxillary Ridge Augmentation Using Autogenous Bone Blocks With and Without Collagen Membranes: A Randomized Controlled Trial. Clin Oral Implants Res. 2025 Nov 3. doi: 10.1111/clr.70059. Online ahead of print. PMID 41184218